CLINICAL TRIAL: NCT00027404
Title: Fluoxetine vs Placebo in Adult Autistic Disorder
Brief Title: Study of Fluoxetine in Adults With Autistic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FD-R-2026-01; FD-R-002026-01
Record Dates: First submitted 2001-12-05; First posted 2001-12-07 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2002-11

CONDITIONS: Autistic Disorder
Keywords: Adult, Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Fluoxetine

INTERVENTIONS:
Drug: Fluoxetine

SUMMARY:
This is a study to determine the effect of fluoxetine in the treatment of adult autism and on functional ability and behavior associated with autism. Evidence suggests abnormal serotonin function in autism. Fluoxetine is a selective inhibitor of the serotonin transporter.

DETAILED DESCRIPTION:
Eligible patients will undergo comprehensive evaluation. Informants familiar with the patient will also provide information. Patients will be randomized to receive treatment or placebo. During the 12-week treatment there will be weekly monitoring for the first 4 weeks and biweekly monitoring for the next 8 weeks. The drug dosage will be increased each week as tolerated by the patient. Serum levels of fluoxetine and norfluoxetine will be documented at Week 12.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
Inclusion criteria:

* Meets DSM-IV and ADI criteria for autistic disorder
* Patients must use effective contraception
* Negative pregnancy test
* Clinical Global Impression-Severity Scale for Autistic Disorder (CGI-AD) score of 4

Exclusion criteria:

* Pregnant or nursing
* Prior or concurrent history of mental disorders, including schizophrenia, schizoaffective disorder, organic mental disorders, or bipolar disorders
* Concurrent depression determined by DSM-IV diagnosis
* Serious suicidal risk
* Active seizure disorder within the past 2 years
* Clinically significant or unstable medical illness, including hematopoietic or cardiovascular disease
* Any organic or systemic disease
* Any geographical condition that would preclude study compliance
* Prior or concurrent gastrointestinal, liver, or kidney disease
* Any other concurrent condition that interferes with the absorption, distribution, metabolism, or excretion of drugs
* Prior or concurrent cerebrovascular disease or brain trauma
* Prior or concurrent clinically significant unstable endocrine disorder, such as hypo- or hyperthyroidism
* Prior or concurrent malignancy
* Clinically significant abnormalities on EKG, laboratory tests, or physical exam
* Requirement for ECT or any other psychotropic medication
* Inability to tolerate taper from psychoactive medication
* History of hypersensitivity or severe side effects associated with the use of fluoxitine or other serotonin reuptake inhibitors
* Treatment with any drug known to have a well-defined potential for toxicity to a major organ within the past 30 days
* Concurrent terfenadine (Seldane) or astemizole (Hismanal)
* Prior treatment with fluoxetine of 40 mg/day for 6 weeks
* Prior electroconvulsive therapy within the past 3 months
* Prior investigational drug use within the past 30 days
* Prior Monoamine oxidase inhibitor use within the past 14 days
* Prior long-acting phenothiazines within the past 6 weeks
* Prior psychotropic drugs within the past 7 days
* Prior fluoxetine within the past 6 weeks
* Requirement for any therapeutic intervention that would confound study evaluation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2001-09; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hollander, MD, Principal Investigator — Mount Sinai School of Medicine New York, New York, United States
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States